CLINICAL TRIAL: NCT01724801
Title: Phase III Study of Icotinib Treat the Patient With Brain Metastasis EGFR-mutant Non Small Cell Lung Cancer Comparing With Whole Brain Radiotherapy
Brief Title: Icotinib or Whole Brain Irradiation in EGFR-mutant Lung Cancer
Acronym: BRAIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Guangdong Association of Clinical Trials (Other)
Collaborators: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTONG1201
Record Dates: First submitted 2012-10-14; First posted 2012-11-12 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Brain Metastasis; Non Small Cell Lung Cancer
Keywords: EGFR mutant
MeSH Terms: conditions — Brain Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — icotinib

ARMS (2):
- icotinib (Experimental): icotinib administered orally at a dose of 125 mg 3 times daily
  Interventions: Drug: Icotinib
- Whole brain irradiation (Active Comparator): Whole brain irradiation 30Gy/3Gy/10 fractions plus concurrent or sequential chemotherapy for 4-6 cycles
  Interventions: Radiation: whole brain radiation(WBI)

INTERVENTIONS:
Radiation: whole brain radiation(WBI) — WBI (30Gy/3Gy/10 fractions) plus concurrent or sequential chemotherapy for 4-6 cycles
  Arms: Whole brain irradiation
Drug: Icotinib — administered orally at a dose of 125 mg 3 times daily
  Arms: icotinib

SUMMARY:
EGFR-TKI is good for the patients with EGFR-mutant non-small cell lung cancer.We design this clinical trail to confirm if the efficacy of Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor(EGFR-TKI )(ICOTINIB) is better than whole brain irradiation for the patient with EGFR-mutant non-small cell lung cancer.

DETAILED DESCRIPTION:
no available

ELIGIBILITY:
Inclusion Criteria:

Patient who was confirmed stage IV NSCLC with EGFR activating mutation and brain metastases by pathologic histology or cytology.

Patient who brain metastases was shown in MRI or CT scan. Brain metastases lesions should be more than 3.The diameter among these lesions should be more than 1 centimeter.

Males or females aged ≥18 years, < 75 years. Eastern Cooperative Oncology Group(ECOG) performance status 0-1. Life expectancy ≥12 weeks. The therapy of surgery,chemotherapy,radiotherapy that the patients were ever received should be more than 2 weeks ago.The patient had recovered from the treatment.

Males and females should be contraceptive during the period of the trial until 8 weeks after the last administration of icotinib.

Able to comply with the required protocol and follow-up procedures, and able to receive oral medications.

Written informed consent provided.

Exclusion Criteria:

Patient was received irradiation of brain. Patient with meningeal metastases were confirmed by MRI or cytology test of cerebrospinal fluid.

Patient is received the treatment of Phenytoin, carbamazepine, rifampicin, phenobarbital, or St. John's Wort.

Patient was received EGFR Tyrosine Kinase Inhibitor or EGFR monoclonal antibody.

Interstitial pneumonia.Pericardial effusion, pleural effusion is uncontrolled .

Any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within the previous year, serious cardiac arrhythmia requiring medication, hepatic, renal, or metabolic disease).

Any significant ophthalmologic abnormality ,especially severe dry eye syndrome ,keratoconjunctivitis sicca,Sjogren syndrome,severe exposure keratitis or any other disorder likely to increase the risk of corneal epithelial lesions.

Lack of physical integrity of the upper gastrointestinal tract, or malabsorption syndrome, or inability to take oral medication, or have active peptic ulcer disease.

Female subjects should not be pregnant or breast-feeding. Adequate hematological function: Absolute neutrophil count (ANC) ≥1.5 x 109/L, and Platelet count ≥100 x 109/L.

Adequate renal function: Serum creatinine ≤ 1.5 x ULN, or ≥ 50 ml/min. Adequate liver function :Total bilirubin £ 1.5 x upper limit of normal (ULN) and Alanine Aminotransferase (ALT )and Aspartate Aminotransferase (AST )< 2.5 x ULN in the absence of liver metastases, or < 5 x ULN in case of liver metastases.

The symptoms of increased intracranial pressure are uncontrolled after dehydration and cortisone treatment.

Patient need increase irradiation dose after routine irradiation(30GY/10f/2w) Patient should treat extra cranial lesions first. Patient assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2012-10-14; Primary Completion 2015-06-30 (Actual); Study Completion 2016-09-14 (Actual)

PRIMARY OUTCOMES:
iPFS | 18 months
  intracranial progression-free survival

SECONDARY OUTCOMES:
progress-free survival (PFS) | up to 16 months
  progress-free survival
time of controlling brain metastasis symptom | 18months
  time of controlling brain metastasis symptom
Response rate of brain metastasis | 12months
  Response rate of brain metastasis
Cognitive function | 18months
  Cognitive function
overall survival(OS) | 24months
  overall survival(OS)

OTHER OUTCOMES:
Toxicity | 24months
  adverse events(according to CTC4.0)

CONTACTS AND LOCATIONS:
Overall Officials: Jinji Yang, MD, Study Director — Guangdong Provincial People's Hospital
Locations (2):
- China (2):
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Guangdong Lung Cancer Institute, Guangdong General Hospital, Guangdong Academy of Medical Sciences, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yang JJ, Zhou C, Huang Y, Feng J, Lu S, Song Y, Huang C, Wu G, Zhang L, Cheng Y, Hu C, Chen G, Zhang L, Liu X, Yan HH, Tan FL, Zhong W, Wu YL. Icotinib versus whole-brain irradiation in patients with EGFR-mutant non-small-cell lung cancer and multiple brain metastases (BRAIN): a multicentre, phase 3, open-label, parallel, randomised controlled trial. Lancet Respir Med. 2017 Sep;5(9):707-716. doi: 10.1016/S2213-2600(17)30262-X. Epub 2017 Jul 19. PMID 28734822